CLINICAL TRIAL: NCT06386627
Title: Study of the Mechanisms of Visual-motor Transformation to Search for Neurophysiological Markers of Changes in the Functions of Cortical Motor Circuits in Patients With Neurological Disorders, and Development of Technologies for Their Rehabilitation.
Brief Title: Study of Neurophysiological Markers of Motor Recovery in Post-stroke Patients.
Status: Completed | Type: Observational
Sponsor: Skolkovo Institute of Science and Technology (Other)
Collaborators: Federal center of brain research and neurotechnologies, FMBA, Moscow, Russia (Unknown)
Responsible Party: Sponsor
Other Study IDs: Skoltech-CNBR3; 21-75-30024 (Other Grant/Funding Number: Russian Science Foundation)
Record Dates: First submitted 2024-04-23; First posted 2024-04-26 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Stroke
Keywords: stroke; hemiparesis; motor cortex; restoration of motor functions; upper limbs
MeSH Terms: conditions — Stroke; Paresis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Post-stroke persons
  Interventions: Diagnostic Test: Stimulus response task; Diagnostic Test: Transcranial magnetic stimulation
- Healthy volunteers
  Interventions: Diagnostic Test: Stimulus response task

INTERVENTIONS:
Diagnostic Test: Stimulus response task — Participants were tasked with performing a finger extension exercise that required pressing buttons in response to visual stimuli. In cases where physical movement was not possible, participants were instructed to imagine performing the task while focusing on their fingers.
Diagnostic Test: Transcranial magnetic stimulation — Transcranial magnetic stimulation to assess the integrity of corticospinal connections
  Groups: Post-stroke persons

SUMMARY:
The aim of the study was to explore potential pathways for recovery and adaptation of neural pathways after stroke by examining electrical activity of the brain cortex and cortico-spinal excitability using transcranial magnetic stimulation in people with motor impairment after stroke. Participants in the study performed a simple stimulus-response task with a healthy and a paralysed limb several times at different stages of basic rehabilitation. To compare the data, a group of healthy volunteers took part in a similar experiment. Investigators recorded cortical activity using electroencephalography and muscle activity using electromyography. After the stimulus-response task, investigators also carried out a study using transcranial magnetic stimulation to assess the integrity of corticospinal connections.

DETAILED DESCRIPTION:
The study involved 40 participants, half of whom had suffered a stroke with hemiparesis and the other half a control group of healthy volunteers. During the experimental session, the participants have to perform a motor task involving reaction speed. A box with two buttons (right and left) is placed in front of the participant. The participant's hands are placed in the box under the buttons. The experimental task is to press one of the two buttons by extending the fingers in response to a visual stimulus - lamps above the buttons. If the degree of damage to the motor function of one of the participant's limbs does not allow a full button to be pressed, the participants is asked to form an intention for this movement and try to perform it. At the same time, one of the buttons has been designated as a 'target' for the patient, and it is in response to its highlighting that a movement is to be performed. The second button is 'non-target'. Its highlighting should be ignored. Throughout the session, each of the buttons was designated as a target several times.

Throughout the session, the electroencephalogram (EEG) signal was recorded in 17 electrodes placed on the scalp according to the international "10-10" registration system. The recording was performed with a medical electroencephalograph NVX-36 ("Medical Computer Systems", Zelenograd, Russia). Electromyographic (EMG) activity of the flexor digitorum superficialis muscles of both hands was also recorded using surface electrodes. The EMG is recorded with the same amplifier as the EEG signal (NVX-36). The participant takes part in the test within 2 weeks. There were two sessions (at the beginning of rehabilitation and before discharge). Each session lasts a maximum of one hour.

Before the study, the participants' motor activity was tested using the Action Research Arm Test (ARAT). The EEG data were analysed for markers such as movement-related potentials and movement-related desynchronisation of alpha and beta rhythms. Some participants were also invited to take part in an additional study using transcranial magnetic stimulation to assess the integrity of corticospinal connections.

ELIGIBILITY:
For Healthy Volunteers:

Inclusion Criteria:

1. Availability of signed written informed consent. 3. Absence of somatic and psychiatric diseases (more details in the exclusion criteria) 4. Ability and willingness to comply with the requirements of this protocol.

Exclusion Criteria:

1. The presence of superficial injury of head (S00-S09 International Classification of Diseases 10 (ICD-10).
2. The presence of mental, behavioural disorders (F00-F99 ICD-10).
3. Drug addiction in the past or at the moment.
4. The presence of diseases of the nervous system (G00-G99 ICD-10).
5. . History of intracranial injury (S06 ICD-10) or stroke (I64 ICD-10).
6. The presence of somatoform disorders (F45 ICD-10).
7. Any conditions that, in the opinion of the Investigator, meet the exclusion criteria
8. Presence of electrical and/or metallic implants or stimulants in the body (eg, implanted deep brain stimulation devices, pacemakers, hearing aids and cochlear implants, intracranial metal implants).
9. Pregnancy
10. The presence of malignant neoplasms (C00-C97 ICD-10).

For stroke patients:

Inclusion Criteria:

1. Signed written informed consent.
2. People after the first acute cerebrovascular accident (CVA), early or late rehabilitation period.
3. The level of severity of paresis of the upper limb from 3 points to 0 (according to a 6-point neurological scale)
4. The minimum visual acuity is not lower than 0.2 on the Sivtsev scale.
5. The ability and willingness of the patient to comply with the requirements of this protocol.
6. Expressed patient motivation for rehabilitation.

Exclusion Criteria:

1. Severe cognitive impairment (<10 points according to the Montreal Cognitive Assessment Scale).
2. Hamilton score above 18 points.
3. The score on the Rankin scale is above 4 points.
4. Associated neurological disorders that cause decreased muscle strength or increased muscle tone in the upper limbs (eg, cerebral palsy, brain damage from trauma) or stiffness (eg, Parkinson's disease, contracture).
5. Late stages of arthritis or clinically significant limitation of passive range of motion in any of the joints studied in the study due to other reasons.
6. The absence of a part of the upper limb due to amputation caused by various reasons.
7. Any medical condition, including mental illness or epilepsy, that may affect the interpretation of study results, study conduct, or patient safety.
8. Alcohol abuse, medical marijuana use, or recreational drug use in the 12 months prior to Visit 1.
9. Use of experimental drugs or medical devices within 30 days prior to Visit 1.
10. Lack of ability to follow study procedures, in the opinion of the investigator.
11. The severity of the patient's condition according to the neurological or somatic status, which does not allow full rehabilitation.
12. Severe visual disturbances, minimal visual acuity less than 0.2 Sivtsev visual acuity table.
13. Unstable angina and/or heart attack within the previous month
14. Repeated stroke.
15. Severe unilateral spatial neglect.
16. Uncontrolled arterial hypertension
17. Ataxia
18. All forms of epilepsy

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing rehabilitation at the Federal center of brain research and neurotechnologies, FMBA, Moscow, Russia.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Atypical shape of lateralized readiness potential | 15 days
  Shape and scalp-distribution of the lateralized pre-motor cortical potentials in post-stroke participants demonstrated bilateral involvement of primary motor cortex, indicating role of healthy hemisphere in the control of impaired limb movements.

SECONDARY OUTCOMES:
Absent of ipsilateral muscles contraction in response to primary motor cortex stimulation in both hemispheres | 1 day
  Transcranial magnetic stimulation did not show increased activity of ipsilateral projections. from intact hemisphere motor cortex to paralyzed limb

CONTACTS AND LOCATIONS:
Locations (1):
- Skolkovo Institute of Science and Technology (Skoltech), Moscow, Russia